CLINICAL TRIAL: NCT02620787
Title: Comparative Assessment of Tedizolid Tissue Penetration and Pharmacokinetic Profile Between Diabetic Patients With Wound Infections and Healthy Volunteers Via In Vivo Microdialysis
Brief Title: Tedizolid Tissue Penetration in Diabetic Patients With Wound Infections and Healthy Volunteers Via In Vivo Microdialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Nicolau-53466
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Wound Infection; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus; Wound Infection | interventions — tedizolid; tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic Wound Infection (Experimental): Participants with a documented medical history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours following the last dose (e.g., 48-72 hours).
  Interventions: Drug: Tedizolid; Procedure: Microdialysis Catheter Insertion
- Healthy Volunteers (Active Comparator): Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours following the last dose (e.g., 48-72 hours).
  Interventions: Drug: Tedizolid; Procedure: Microdialysis Catheter Insertion

INTERVENTIONS:
Drug: Tedizolid
  Other Names: Sivextro
Procedure: Microdialysis Catheter Insertion — A 20 kila-Dalton microdialysis probe (63 MD catheter; MDialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous tissue at the margin of the wound (patient group) or in the thigh tissue (healthy volunteers). The probe will be left in place for the final dose and all tissue sampling procedures thereafter. This probe is perfused with a physiologic solution to collect interstitial fluid samples. The probe will then be removed after completion of sample collection.

SUMMARY:
This study will determine the tissue penetration of tedizolid (Sivextro, Merck & Co.), a novel oxazolidinone antibiotic, into the extracellular, interstitial fluid of soft tissue in diabetic patients with lower limb wound infections. Penetration will be compared with a group of healthy volunteer control participants.

DETAILED DESCRIPTION:
This study will enroll 10 patients with diabetes who are admitted with a lower limb wound infection and 6 healthy volunteer control participants. The study will take place in an inpatient unit at Hartford Hospital for all patients and in the Clinical Research Center at Hartford Hospital for all healthy volunteers. All participants will receive 3 to 6 doses of oral tedizolid 200mg once daily. A microdialysis probe (Mdialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous soft tissue near the margin of the wound (patients) or in the thigh (healthy volunteers). The microdialysis probe is perfused with lactated Ringer's solution and samples are collected for the 24 hours following the final dose (i.e., 48-72 hours). A peripheral intravenous catheter will be inserted into an arm vein to collect blood samples simultaneously with microdialysis samples. Concentrations in tissue are compared with blood to determine percent penetration.

ELIGIBILITY:
Inclusion Criteria:

* Experimental: Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb
* Active Comparator: Healthy Adult Volunteer

Exclusion Criteria:

All Participants:

* Less than 18 years of age
* History of hypersensitivity to tedizolid or linezolid
* History of hypersensitivity to lidocaine or lidocaine derivatives
* Pregnant or breastfeeding
* Presence of anemia, thrombocytopenia, or leukopenia as defined by hematocrit, platelet, or white blood cell count < 75% of the lower limit of normal
* Concomitant receipt of linezolid
* Any other reason felt by the investigator to potentially affect the outcomes of the study

Experimental Group Only:

* No palpable pedal pulses present
* Participants likely to require multiple surgical interventions during the study period, which therefore could affect placement of the microdialysis catheter

Active Comparator Group Only:

* Positive urine drug screen (cocaine, tetrahydrocannabinol, opiates, benzodiazepines, and amphetamines).
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalence of 5 cigarettes per day.
* Use of prescription or nonprescription drugs, vitamins, or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, with the exception of acetaminophen at doses of ≤ 1 g/day. Herbal supplements, hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing intrauterine devices (IUDs), postcoital contraceptive methods), and hormone replacement therapy must be discontinued at least 14 days prior to the first dose of study medication. Depo-Provera® must be discontinued at least 6 months prior to the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Nicolau, PharmD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Wound Infection: Participants with a documented medical history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours.
- Healthy Volunteers: Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours.
Period: Overall Study
Arm/Group | Diabetic Wound Infection | Healthy Volunteers
Started | 12 | 6
Completed | 10 | 6
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Eligibility Criteria Not Met | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diabetic Wound Infection: Participants with a documented medical history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours.
  Tedizolid
  Microdialysis Catheter Insertion: A 20 kila-Dalton microdialysis probe (63 MD catheter; MDialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous tissue at the margin of the wound (patient group) or in the thigh tissue (healthy volunteers). The probe will be left in place for the final dose and all tissue sampling procedures thereafter. This probe is perfused with a physiologic solution to collect interstitial fluid samples. The probe will then be removed after completion of sample collection.
- Healthy Volunteers: Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive 3 to 6 doses of oral tedizolid 200mg once daily, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 24 hours.
  Tedizolid
  Microdialysis Catheter Insertion: A 20 kila-Dalton microdialysis probe (63 MD catheter; MDialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous tissue at the margin of the wound (patient group) or in the thigh tissue (healthy volunteers). The probe will be left in place for the final dose and all tissue sampling procedures thereafter. This probe is perfused with a physiologic solution to collect interstitial fluid samples. The probe will then be removed after completion of sample collection.
- Total: Total of all reporting groups
Arm/Group | Diabetic Wound Infection | Healthy Volunteers | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (17) | 33 (9) | 44 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 8
  Not Hispanic or Latino | 2 | 6 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 5 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (6.3) | 28.5 (5.4) | 30.4 (6.0)
Weight [Mean (Standard Deviation); unit: kg] | 89.4 (21) | 79.5 (17.9) | 85.7 (19.9)
Height [Mean (Standard Deviation); unit: inches] | 66.6 (5.0) | 65.7 (4.5) | 66.3 (4.7)
Albumin [Mean (Standard Deviation); unit: g/dL] | 3.1 (0.4) | 4.6 (0.3) | 3.6 (0.8)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.2) | 0.9 (0.1) | 0.9 (0.2)
Creatinine clearance [Mean (Standard Deviation); unit: mg/ml] | 90.4 (31.9) | 101.5 (26.6) | 94.6 (29.6)
PEDIS Grade [Count of Participants; unit: Participants] — Grade 2 Presence of ≥2 manifestations of inflammation (purulence, or erythema, pain, tenderness, warmth, or induration), but any cellulitis/erythema ≤2 cm around the ulcer, and infection is limited to the skin or superficial subcutaneous tissues; no other local complications or systemic illness
  Grade 3 Infection (as above) in a participant systemically well, metabolically stable but has ≥1 of the following: cellulitis extending >2 cm, lymphangitic streaking, spread beneath superficial fascia, deep-tissue abscess, gangrene, and involvement of muscle, tendon, joint or bone Population: Only patient participants were analysed for PEDIS grade. Healthy volunteers (i.e. non diabetics) did not exibit wound infections.
  Participants
    number analyzed (Participants) | 10 | 0 | 10
    Grade 2 | 1 |  | 1
    Grade 3 | 9 |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Tedizolid Tissue Penetration
Description: The ratio of tedizolid tissue concentrations to blood concentrations following the final tedizolid dose
Time Frame: 48-72 hours
Population: One volunteer and one patient participant were excluded due to low concentrations
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Diabetic Wound Infection | Healthy Volunteers
Number analyzed (Participants) | 9 | 5
ratio | 0.98 (0.43) | 0.82 (0.08)

2. Secondary Outcome: Tedizolid Area Under the Curve (AUC) in Tissue
Description: The area under the drug concentration-time curve (AUC) in tissue reflects the actual tissue exposure to drug after administration of a dose of the drug and is expressed in mg*h/L.
  Venous blood was obtained via peripheral intravenous catheter at 48 hours from the start of the first dose (i.e., immediately before administration of the 3rd dose), and at 49, 50, 50.5, 51, 51.5, 52, 54, 56, 60, 64 and 72 hours.
  Dialysate samples of 120μL were collected in 200µL microvials simultaneously with plasma at 48, 49, 50, 51, 52, 53, 54, 55, 56, 57, 58, 59, 60, 64, 68 and 72 hours following administration of the first dose.
Time Frame: 48-72 hours
Population: One volunteer and one patient participant were excluded due to low concentrations
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Diabetic Wound Infection | Healthy Volunteers
Number analyzed (Participants) | 9 | 5
mg*h/L | 3.44 (1.50) | 5.20 (1.61)

3. Secondary Outcome: Tedizolid AUC in Plasma
Description: The area under the plasma drug concentration-time curve (AUC) reflects the actual plasma exposure to drug after administration of a dose of the drug and is expressed in mg*h/L
Time Frame: 48-72 hours
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Diabetic Wound Infection | Healthy Volunteers
Number analyzed (Participants) | 10 | 6
mg*h/L | 18.47 (9.70) | 28.71 (9.58)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a 76 hour window, from the start of first tedizolid dose (0 hour) to the end of blood/dialysate sampling (72 hours), plus a 4 hour observation window after the last sample was collected for subjects who received at least one dose of tedizolid. Note. In the diabetic wound infection group, 12 subjects were enrolled, but 11 received at least one dose. Therefore, the denominator is different from what is listed in the participant flow.
Description: Adverse event: any pathologic or unintended change in the structure, function, or chemistry associated with the use of the study drug, whether or not considered drug related:
  MILD - present, but easily tolerated MODERATE - discomfort that interferes with usual activities SEVERE - incapacitating, inability to do usual activities
  A serious adverse event will be defined as any which results in death or is immediately life-threatening, requires in-participant hospitalization.
Arm/Group | Diabetic Wound Infection | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6
Other Adverse Events (participants affected / at risk) | 2/11 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diabetic Wound Infection (N=11) | Healthy Volunteers (N=6)
Headache (Nervous system disorders) | 0 | 3
Hypothermia (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02620787/Prot_SAP_000.pdf